CLINICAL TRIAL: NCT03688061
Title: A Phase-I Dose-Escalation Study to Evaluate the Safety and Immunogenicity of Prime-Boost Immunisations With Candidate HCV Vaccines, ChAd3-hliNSMut and MVA-hliNSMut in Healthy Volunteers and Patients Previously Chronically Infected With HCV
Brief Title: Class II Invariant Chain HCV Vaccine Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Oxford University Hospitals NHS Trust (Other); ReiThera Srl (Industry); European Commission (Other); GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: PEACHI-03; 2016-000983-41 (EudraCT Number)
Record Dates: First submitted 2018-09-19; First posted 2018-09-27 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2018-09

CONDITIONS: Hepatitis C
Keywords: Hepatitis; Vaccine; Adenoviral-vector; human invariant chain
MeSH Terms: conditions — Hepatitis C; Hepatitis

STUDY DESIGN:
Intervention Model Description: Each group will be sequentially recruited over a period of two months to allow for safety review.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group 1 (low dose/healthy volunteers) (Experimental): 5 healthy volunteers receiving 1 dose ChAd3-hliNSmut (5x10*9 vp) IM at week 0 and 1 dose of MVA-hliNSmut (5 X10*7 pfu) IM at week 8
  Interventions: Biological: ChAd3-hliNSmut; Biological: MVA-hliNSmut
- Group 2 (higher dose/healthy volunteers) (Experimental): 10 healthy volunteers receiving 1 dose ChAd3-hliNSmut (2.5 x10*10 vp) IM at week 0 and 1 dose of MVA-hliNSmut (2 X 10*8 pfu) IM at week 8
  Interventions: Biological: ChAd3-hliNSmut; Biological: MVA-hliNSmut
- Group 3 (higher dose/HCV cured volunteers) (Experimental): 10 DAA treated volunteers (previously HCV positive) receiving 1 dose ChAd3-hliNSmut (2.5 x10*10 vp) IM at week 0 and 1 dose of MVA-hliNSmut (2 X10*8 pfu) IM at week 8
  Interventions: Biological: ChAd3-hliNSmut; Biological: MVA-hliNSmut

INTERVENTIONS:
Biological: ChAd3-hliNSmut — Attenuated chimpanzee adenovirus (ChAd) vectored vaccine against HCV
Biological: MVA-hliNSmut — Modified Vaccinia Ankara (MVA) vectored vaccine against HCV

SUMMARY:
The study is aimed at assessing the safety and immunogenicity of HCV prime-boost vaccinations ChAd3-hliNSmut and MVA-hliNSmut, administered intramuscularly in healthy volunteers and DAA treated patients.

DETAILED DESCRIPTION:
Hepatitis C currently infects more than 180 million people worldwide and is associated with the development of liver cancer, liver failure and liver cirrhosis. Although drug treatments are available these are expensive and prolonged. Furthermore patients often only present to health care professionals at late stages when liver disease has already progressed. Therefore, vaccination remains the optimal method of preventing infection. To date this has proved extremely difficult due to the enormous variation in HCV strains around the world.

Researchers at the University of Oxford in collaboration with industry, have developed novel candidate vaccines against HCV ('NSmut'). These vaccines have been inserted into the carrier viruses Chimpanzee Adenovirus (ChAd) and modified vaccinia virus Ankara (MVA), both of which have excellent safety records. These vaccines have been given to hundreds of healthy volunteers and are now being tested for effectiveness.

In this study we are hoping to increase the immune response against the HCV virus. We will do this by inserting a gene in the vaccine (class-II invariant gene). In animal studies, this approach has been shown to be safe and to significantly to enhance the immune response against HCV.

During this study 15 healthy adults and 10 volunteers who were previously treated for HCV infection, aged 18-65 years, will receive either two intramuscular injections over a period of two months. All participants will be followed up for a further 6 months (12 visits in total) and will be asked to give a blood sample at each clinic visit.

The aims of the study are to assess the safety of the vaccine and to see if the vaccine can induce a strong immune response against the hepatitis C Virus.

ELIGIBILITY:
Inclusion Criteria:

* Aged at least 18 years on the day of screening and no greater than 65 years on the day of the first vaccination
* Resident in or easy access to the trial site for the duration of the study
* Available for follow-up for the planned duration of the study
* Able and willing (in the CI's opinion) to comply with all study requirements
* Willing to allow the investigators to discuss the volunteer's medical history with their General Practitioner
* For heterosexual females, willingness to practice continuous effective contraception from screening until 4 months after the last immunisation
* All female volunteers must be willing to undergo urine pregnancy tests at the time points specified in the Schedule of Procedures and must have a negative pregnancy test on the day(s) of vaccination
* For sexually active men, willingness to use condoms from screening until 4 months after the last vaccination
* Agreement to refrain from blood donation during the course of the study
* In the opinion of the Chief Investigator or designee, the volunteer has understood the information provided. Written informed consent must be given before any study-related procedures are performed
* Willing to undergo HCV and HIV testing, counselling and receive test results

Specific for Groups 1 and 2:

• Healthy males or females, as assessed by medical history, physical examination and laboratory tests

Specific for Group 3:

* A previous diagnosis of chronic HCV infection (any HCV genotype) successfully treated with all oral DAA therapy.
* Minimum duration of six months between last dose of DAA treatment and planned vaccination date
* SVR 12 following last DAA treatment course
* Fibroscan score of <12.5kPa within 6 months of screening.

Exclusion Criteria:

* Participation in another research study involving an investigational product in the 30 days preceding enrolment, or planned used during the study period
* Prior receipt of a recombinant simian adenoviral vaccine
* Receipt of any investigational HCV vaccine within the last 6 years
* Administration of immunoglobulins and/or any blood products within the last three months preceding the planned administration of the vaccine candidate
* Receipt of live attenuated vaccine within the previous 60 days or planned receipt within 60 days after vaccination with the IMP
* Receipt of other vaccine, including influenza vaccine, within the previous 14 days or planned receipt within 14 days after vaccination with the IMP
* Any confirmed or suspected immunosuppressive or immunodeficient state, including HIV infection; asplenia; recurrent, severe infections and chronic (more than 14 days) immunosuppressive medication within the last 6 months (inhaled and topical steroids are allowed)
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine
* Any history of anaphylaxis in reaction to vaccination
* Pregnancy, lactation or willingness/intention to become pregnant during the study
* Personal history of autoimmune disease
* History of major autoimmune disease in first degree relative, e.g. Type 1 diabetes, Graves' Disease, Systemic Lupus Erythematosus (SLE) or Spondyloarthropathy (AS).
* HLA type B27 positive individuals
* History of cancer (except basal cell carcinoma of the skin and cervical carcinoma in situ)
* History of serious psychiatric condition
* Any other serious chronic illness requiring hospital specialist supervision
* Suspected or known current alcohol abuse as defined by an alcohol intake of greater than 42 units every week
* Suspected or known current injecting drug use
* Seropositive for hepatitis B surface antigen (HBsAg)
* Any clinically significant acute or chronic medical condition that is considered unstable/progressive, or in the opinion of the Chief Investigator, may either put the volunteer at risk because of participation in the study, or may influence the result of the study, or the volunteer's ability to participate in the study
* Any clinically significant abnormal finding on screening biochemistry or haematology blood test or urinalysis
* Any other finding which in the opinion of the investigators would significantly increase the risk of having an adverse outcome from participating in the protocol
* Vulnerable subjects (according to ICH GCP)

Specific for groups 1 and 2:

* Previous HCV infection
* Reported current or previous high-risk behaviour for HCV infection (including IVDU)
* Seropositive for hepatitis C virus (antibodies to HCV) at screening

Specific for group 3:

* Reported current high-risk behaviour for HCV infection (previous IVDU is not an exclusion criteria for this group)
* HCV RNA positive following DAA treatment
* Cirrhosis or severe fibrosis (Ishak 5 or 6) as previously defined by any of the following:

  * Radiological findings on CT, MR or USS
  * Abnormal biochemical parameters (PT, albumin and bilirubin)
  * clinical signs of liver decompensation (ascites, varices, encephalopathy)
  * Ishak score 5 on liver biopsy
  * Fibroscan at any time point in the past >12.5kPa

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2017-12-04 (Actual); Primary Completion 2019-08-04 (Actual); Study Completion 2022-08-04 (Actual)

PRIMARY OUTCOMES:
Proportion of volunteers who develop a grade 3 local and systemic reactions | Actively collected throughout the study until 6 months after the last vaccination
  To evaluate the safety of administering HCV prime-boost vaccinations, ChAd3-hliNSmut and MVA-hilNSmut intramuscularly in healthy volunteers and DAA treated volunteers that were previously infected with HCV

SECONDARY OUTCOMES:
Proportion of volunteers who develop T cell responses to HCV epitopes, as determined by INF-gamma ELISpot assay | Actively collected throughout the study until 6 months after the last vaccination
  To assess the cellular immune response generated by HCV prime-boost vaccinations, ChAd3-hliNSmut and MVA-hliNSmut administered intramuscularly to healthy volunteers and DAA treated volunteers that were previously infected with HCV

CONTACTS AND LOCATIONS:
Overall Officials: Eleanor Barnes, Professor, Study Chair — University of Oxford; Lucy Dorrell, Professor, Principal Investigator — University of Oxford
Locations (2):
- United Kingdom (2):
  - Centre for Cinical Vaccinology and Tropical Medicine, Univeristy of Oxford, Oxford, Oxfordshire
  - Hepatology Clinical Trial Unit, John Radcliffe Hospital, Oxford, Oxfordshire

IPD SHARING:
Plan to Share IPD: Undecided